CLINICAL TRIAL: NCT04711447
Title: Effect of Inhibitory Kinesio-tape of the Upper Trapezius on Lower Trapezius Muscle Excitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trisha Scribbans (Other)
Responsible Party: Sponsor-Investigator, Trisha Scribbans, Associate Professor, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HS22668 (E2019:019)
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Scapular Dyskinesis
Keywords: kinesio tape (KT); Shoulder; upper trapezius; lower trapezius
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no-tape, experimental KT, sham KT (Other): Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both an experimental-KT (E-KT) and sham-KT (S-KT) condition.
  Interventions: Device: kinesio-tape
- no-tape, sham KT, experimental KT (Other): Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both a sham-KT (S-KT) condition and experimental-KT (E-KT).
  Interventions: Device: kinesio-tape

INTERVENTIONS:
Device: kinesio-tape — Twenty-two individuals with healthy shoulders completed 10 repetitions of an arm elevation task during three taping conditions (no-tape, experimental KT, sham KT) and 2 loading conditions (no-load and loaded).

SUMMARY:
Shoulder pain increases excitation (or activity) of the upper trapezius (UT) and reduces excitation in lower trapezius (LT). Despite inconclusive evidence, kinesio-tape (KT) is often used to modify muscular excitation within the UT and/or LT to help correct alterations in scapular position and motion associated with shoulder pain/injury. The objectives of the current study were to determine if: 1) inhibitory KT to the UT acutely increases muscle excitation (whole-muscle and spatial distribution) within the LT in healthy individuals; and 2) if loading the limb alters the magnitude of change in muscle excitation of the LT. We hypothesize that: 1) inhibitory KT application to the UT will immediately increase whole-muscle LT excitation, and result in an inferior shift in the distribution of excitation within the LT compared to no tape and sham-KT tape conditions; and 2) the magnitude of immediate increase in LT excitation with KT would be greater in the loaded condition. A repeated-measures, crossover design was used to determine the impact of KT applied to UT and load on muscle excitation of the LT. Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. A baseline trial (no KT; N-KT) was performed first, followed by both an experimental-KT (E-KT) and sham-KT (S-KT) condition. The order of the E-KT and S-KT conditions were randomized and the order was counterbalanced. Testing for each tape condition lasted approximately 10-minutes for a total of 45-minutes per participant including screening, EMG set-up and clean-up. KT was applied to the UT and muscle excitation (EMG amplitude) was measured in the LT using one single 32-grid high-density surface electromyography (HD-sEMG) electrode during a repeated arm elevation task.

ELIGIBILITY:
Inclusion Criteria:

* right-handed individuals
* no current shoulder pain or pathology in the shoulder, neck, back.

Exclusion Criteria:

* recent history (<6 months) of injury or orthopedic disorder of the shoulder, upper back or neck (e.g. rotator cuff tears, disc pathologies, etc.)
* neurological or musculoskeletal disorder (e.g. epilepsy, multiple sclerosis, etc.)
* current pain in the shoulder, upper back or neck
* previous allergies or skin irritation to adhesives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Scribbans, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants excluded due to not meeting inclusion criteria.
Period: Overall Study
Arm/Group | No-tape, Experimental KT, Sham KT | No-tape, Sham KT, Experimental KT
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No-tape, Experimental KT, Sham KT: Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both an experimental-KT (E-KT) and sham-KT (S-KT) condition.
  kinesio-tape: Twenty-one individuals with healthy shoulders completed 10 repetitions of an arm elevation task during three taping conditions (no-tape, experimental KT, sham KT) and 2 loading conditions (no-load and loaded).
- No-tape, Sham KT, Experimental KT: Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both a sham-KT (S-KT) condition and experimental-KT (E-KT).
  kinesio-tape: Twenty-one individuals with healthy shoulders completed 10 repetitions of an arm elevation task during three taping conditions (no-tape, experimental KT, sham KT) and 2 loading conditions (no-load and loaded).
- Total: Total of all reporting groups
Arm/Group | No-tape, Experimental KT, Sham KT | No-tape, Sham KT, Experimental KT | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24 (3) | 24 (3) | 24 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Whole-muscle Activation
Description: RMS measured using high-density EMG electrode grids
Time Frame: Measured during 2nd-9th repetitions of the arm elevation task. Each repetition lasted approximately 1.5 seconds, thus the timeframe was approximately 12 seconds.
Measure: Mean (Standard Deviation); unit: V
Groups:
- No-tape, no Load: Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both an experimental-KT (E-KT) and sham-KT (S-KT) condition.
  kinesio-tape: Twenty-one individuals with healthy shoulders completed 10 repetitions of an arm elevation task during three taping conditions (no-tape, experimental KT, sham KT) and 2 loading conditions (no-load and loaded).
- Sham KT, No-load; Kinesio Tape, No-load; No-tape, With Load; Sham KT, With Load; Kinesio Tape, With Load: Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both a sham-KT (S-KT) condition and experimental-KT (E-KT).
  kinesio-tape: Twenty-one individuals with healthy shoulders completed 10 repetitions of an arm elevation task during three taping conditions (no-tape, experimental KT, sham KT) and 2 loading conditions (no-load and loaded).
Arm/Group | No-tape, no Load | Sham KT, No-load | Kinesio Tape, No-load | No-tape, With Load | Sham KT, With Load | Kinesio Tape, With Load
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
V | .046 (.019) | .043 (.015) | .040 (.018) | .061 (.021) | .065 (.020) | .064 (.026)

2. Secondary Outcome: Spatial Distribution of Muscle Activation
Description: shifts in excitation measured using high-density EMG electrode grids
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Row 1 Baseline; Row 1 Sham; Row 1 KT; Row 2 Baseline; Row 2 Sham; Row 2 KT; Row 3 Baseline; Row 3 Sham; Row 3 kt; Row 4 Baseline; Row 4 Sham; Row 4 kt; Row 5 Baseline; Row 5 Sham; Row 5 KT; Row 6 Baseline; Row 6 Sham; Row 6 KT; Row 7 Baseline; Row 7 Sham; Row 7 KT; Row 8 Baseline; Row 8 Sham; Row 8 KT: Participants were asked to perform a repeated arm elevation task during three different taping conditions: no KT, experimental KT and sham KT. Each taping condition performed the repeated arm elevation task during two loading conditions: no load and loaded with 2.3 kilograms. All six conditions were tested during one visit with the no load condition preceding the loaded condition for each taping condition. This trial consisted of a baseline trial (no KT; N-KT) that was performed first, followed by both an experimental-KT (E-KT) and sham-KT (S-KT) condition.
  kinesio-tape: Twenty-one individuals with healthy shoulders completed 10 repetitions of an arm elevation task during three taping conditions (no-tape, experimental KT, sham KT) and 2 loading conditions (no-load and loaded).
  Individual rows of electrodes were compared during the weighted condition between N-KT, E-KT, and S-KT.
Arm/Group | Row 1 Baseline | Row 1 Sham | Row 1 KT | Row 2 Baseline | Row 2 Sham | Row 2 KT | Row 3 Baseline | Row 3 Sham | Row 3 kt | Row 4 Baseline | Row 4 Sham | Row 4 kt | Row 5 Baseline | Row 5 Sham | Row 5 KT | Row 6 Baseline | Row 6 Sham | Row 6 KT | Row 7 Baseline | Row 7 Sham | Row 7 KT | Row 8 Baseline | Row 8 Sham | Row 8 KT
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
mV | .111 (.05) | .114 (.05) | .111 (.06) | .105 (.04) | .111 (.04) | .109 (.047) | .088 (.03) | .093 (.03) | .093 (.03) | .066 (.02) | .07 (.02) | .07 (.03) | .05 (.02) | .05 (.02) | .05 (.02) | .03 (.01) | .03 (.01) | .04 (.01) | .02 (.01) | .02 (.01) | .03 (.01) | .02 (.01) | .02 (.01) | .02 (.01)

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected.
Description: The use of kinesio-tape is not associated with adverse events. As we did not administer a therapy that would experience adverse events, we did not collect or report adverse events as per the definition of clinicaltrials.gov
Groups:
- Experimental KT: Participants received an upper trapezius inhibitory kinesio-tape tape application that was left on only during the arm elevation task. The upper trapezius was placed in a lengthened position and the tape was applied parallel with the muscle fibres at ~125% tension from original length.
- Sham KT: Participants received an upper trapezius sham kinesio-tape application that was left on only during the arm elevation task. The tape was applied with the participant in resting position (i.e., the muscle was not stretched or shortened) and laid gently parallel with the muscle fibres with no stretch to the tape.
Arm/Group | Experimental KT | Sham KT
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No washout period utilized could lead to compounding effects of the kinesio-tape or sham tape conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT04711447/Prot_SAP_000.pdf